CLINICAL TRIAL: NCT05561946
Title: An Observational Study of Skin Reaction in Infants Using the Owlet Sock OSS 3.0
Status: Completed | Type: Observational
Sponsor: Owlet Baby Care, Inc. (Industry)
Collaborators: Louisiana State University Health Sciences Center Shreveport (Other); University of Utah (Other); Topaz Clinical Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: OWL 2021-01
Record Dates: First submitted 2022-09-19; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Skin Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalized Infants: Hospitalized infants that are planned/scheduled to remain in-house for at least 2 days will wear the sock for a minimum of 48 hours and a maximum of 14 days.
  Interventions: Device: Owlet OSS 3.0
- Healthy Infants: Healthy infants, accompanied by their parent or legal guardian, that are able to stay at a clinical site for 2 days to complete a minimum of 48 hours of monitoring.
  Interventions: Device: Owlet OSS 3.0

INTERVENTIONS:
Device: Owlet OSS 3.0 — The Owlet OSS 3.0 is worn continuously for a minimum of 48 hours and the skin where the device is worn is monitored for any skin injury/irritation

SUMMARY:
This multi-center, open-label, observational study will evaluate possible skin reactions associated with the wearing of the Owlet OSS 3.0 device continuously (except during sensor charging and excessive motion) up to 24 hours per day in a clinical environment.

DETAILED DESCRIPTION:
After an informed consent process, the Owlet OSS 3.0 Sock device will be applied to the foot in accordance with the instructions for use for the device. A research team member, along with any appropriate medical personnel, will perform a baseline examination of the skin to ensure there are no preexisting skin or extremity findings which would interfere with interpretation of subsequent examinations.

A review of the medical record will be performed with the consent process to ensure that vital signs and the cardiorespiratory status of the patient is sufficiently stable for the patient to proceed with study participation. A verbal medical history from the parent may be performed in lieu of a medical record review in healthy subjects.

Subject height and weight, and measurements of the circumference of the subject's ankle and midfoot will be performed at the start of the study and recorded. Sock size will be estimated according to subject weight, per the instructions for use.

The device will be worn by the subject continuously, except during skin assessments, when devices are exchanged, or activities of daily living such as bathing and brief ambulation for toddlers.

A baseline photograph will be taken of the study subject's feet and labeled as right/left, to be kept for reference for future skin exams. Skin examinations will be performed every 4 hours on the foot where the device is placed, including with repositioning. A ±30-minute window on either side of the prescribed time will be acceptable (1 hour total) to comply with the schedule of events.

Repositioning the device to the opposite foot will occur routinely every 8 hours, or sooner if there is evidence of a skin reaction related to device wear. Again, a ±30-minute window on either side of the prescribed time will be acceptable for protocol compliance.

A photograph will be taken of the study subject's feet at baseline prior to application of the Owlet Sock OSS 3.0 device. A photograph of the initial application of the device will also be taken and documented in the study subject's record.

Documentation of the date, time, location, and result of each skin exam will be performed. Photographs of any skin reactions with a severity level of 1-7 will be taken. If any skin reactions are observed, the device will not be placed on the affected foot until the reaction has resolved and returned to baseline. The device will be applied to the unaffected foot while the affected foot reaction resolves. If the skin finding does not resolve within the allowed 8 hour window when the sock must be rotated to the opposite foot, the subject will be withdrawn from study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form by the legal guardian
* Stated willingness of the guardian to adhere to study procedures and availability for the duration of the study
* Anticipated to maintain continuity of study procedures under study team oversight for a minimum of 48 hours duration
* Male or female infants aged 1 month (44 weeks corrected gestational age) to 18 months, with weight between 5 and 30 lbs who will be observed in a hospital pediatric department, or other clinical site

Exclusion Criteria:

* Medical conditions determined by the study subject's physician or site investigator that would prevent their participation
* Presence of any devices or medical equipment that in the opinion of the investigator would interfere with the function of the Owlet device or preclude completion of the protocol
* Patients on vasoactive medications
* Known allergic reactions to nylon, spandex, elastine or polyester film components of the device that will come into contact with skin
* Local skin disease prohibiting wearing of the device

Ages: 44 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants admitted for care and estimated to be in the hospital ward/unit, and healthy infants able to stay at a clinical site with study team oversight for at least 48 hours.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Clinically Important Skin Reactions | From baseline to study completion
  To estimate the incidence of clinically important skin reactions associated with the Owlet Sock OSS 3.0 when instructions for use are followed.

SECONDARY OUTCOMES:
Skin reaction resolution | From onset of observation of skin finding until end of study participation, up to 30 days.
  Measure the time intervals for resolution of a skin finding related to wear of the device.
Estimate the proportion of skin reactions that require medical intervention. | During period of study monitoring, approximately 14 days.
  Categorical determination for need of medical intervention, and description of what type of treatment applied.
Estimate the incidence of any skin reactions, overall and by severity level. | From initiation of study intervention to end of study intervention, approximately 14 days.
  Measurement of total number of skin findings of any type related to device wear.

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Niksch, MD, Study Director — Study Sponsor
Locations (2):
- United States (2):
  - TOPAZ Clinical Research, Apopka, Florida
  - Louisiana State University Health Shreveport, Shreveport, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. MHealth: New Horizons for Health through Mobile Technologies (Global Observatory for Ehealth). 1st ed., World Health Organization, 2011.
- [Background] Dangerfield MI, Ward K, Davidson L, Adamian M. Initial Experience and Usage Patterns With the Owlet Smart Sock Monitor in 47,495 Newborns. Glob Pediatr Health. 2017 Dec 4;4:2333794X17742751. doi: 10.1177/2333794X17742751. eCollection 2017. PMID 29230431
- [Background] Panda SS, Panda M, Das RR, Mohanty PK. Pulse oximeter probe-induced toe injury in a neonate: A rare avoidable injury. J Clin Neonatol 2014;3:240